CLINICAL TRIAL: NCT00891072
Title: A Phase 1 Study of R-(-)-Gossypol (Ascenta's AT-101) in Combination With Paclitaxel and Carboplatin in Solid Tumors
Brief Title: Gossypol, Paclitaxel, and Carboplatin in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03109; 050905; U01CA132194 (NIH); CDR0000640622 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — gossypol acetic acid; Paclitaxel; Taxes; Carboplatin

ARMS (1):
- Treatment (Experimental): Patients receive oral R-(-)-gossypol acetic acid twice daily on days 1-3. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: R-(-)-gossypol acetic acid; Drug: paclitaxel; Drug: carboplatin; Other: pharmacological study

INTERVENTIONS:
Drug: R-(-)-gossypol acetic acid — Given orally
  Other Names: AT-101
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of gossypol when given together with paclitaxel and carboplatin in treating patients with solid tumors that are metastatic or cannot be removed by surgery. Drugs used in chemotherapy, such as gossypol, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gossypol together with paclitaxel and carboplatin may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary end point will be to determine the maximum tolerated dose of AT-101 with paclitaxel and carboplatin.

SECONDARY OBJECTIVES:

I. To describe the toxicities associated with the combination of paclitaxel, carboplatin, and AT-101.

II. To evaluate the human pharmacokinetic disposition of AT-101 in the context of escalating doses.

III. To describe the pharmacokinetics of paclitaxel when given concurrently with AT-101.

IV. To evaluate for evidence of activity for the combination of paclitaxel, carboplatin and AT-101.

OUTLINE: This is a dose-escalation study of R-(-)-gossypol acetic acid.

Patients receive oral R-(-)-gossypol acetic acid twice daily on days 1-3. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic and pharmacodynamic studies by liquid chromatography/mass spectrometry.

After completion of study therapy, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignancy that is metastatic and unresectable and for which standard curative or palliative measures do not exist or are no longer effective; patient may have previously treated or untreated disease
* Patients may have had no more than nine months of previous marrow damaging cytotoxic chemotherapy; examples include but are not limited to: platinum agents cyclophosphamide, ifosfamide, BCNU, and mitomycin C; chemotherapy agents that are non-alkylators such as fluorouracil or taxanes will not be considered marrow damaging chemotherapy; patients must be at least 28 days from last prior chemotherapy or molecular therapy; at least six weeks from last chemotherapy if the regimen included BCNU or mitomycin C; it must be at least 2 weeks from last radiation therapy and less than a total of 30% of the bone marrow receiving radiation dose > 3000 cGy; in addition, patients may not have received previous high-dose therapy requiring hematopoietic stem cell transplantation nor can they have received anti-cancer treatments involving radioactive pharmaceuticals
* Patients with non-Hodgkins lymphoma that is amenable to hematopoietic stem cell transplantation with curative intent may participate only if stem cell transplant is refused or is not indicated
* ECOG performance status =< 2, Karnofsky ≥ 60%
* Life expectancy of greater than 3 months
* Absolute Neutrophil Count ≥ 1,500/uL
* Platelets ≥ 100,000/uL
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) =< 2.5 X institutional ULN
* Creatinine within normal institutional limits OR a measured creatinine clearance by 24 hour urine collection greater than 60 mL/min; a calculated creatinine clearance by Cockcroft-Gault Formula is acceptable in lieu of a measured value
* All Patients must have Measurable or Evaluable Disease per RECIST Criteria
* The effects of AT-101 on the developing human fetus are unknown; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation, and for at least one month following the last dose of AT-101; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with previously treated brain metastases who are clinically and radiographically stable or improved at least four weeks after completion of radiation therapy and are off steroids are eligible; an MRI of the brain or CT scan of the head with contrast must be performed at baseline for patients with history of and/or symptoms suspicious of brain metastases
* Patients must sign informed consent

Exclusion Criteria:

* Treatment with chemotherapy, hormonal agents (except LHRH agonists/antagonists) used for their anti-cancer activity, or biologic response modifiers within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Failure to recover fully (as judged by the investigator) from prior surgical procedures, or failure to recover from adverse events due to agents administered more than 4 weeks earlier
* Concurrent treatment with an investigational agent other than the investigational agent(s) used in this study OR treatment within 4 weeks of study entry with any investigational agent(s) or device(s)
* Any prior use of racemic gossypol or AT-101
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AT-101 or other agents used in study
* Requirement for routine use of hematopoietic growth factors (including granulocyte colony stimulating factor, granulocyte macrophage colony stimulating factor, or interleukin-11) or platelet transfusions to maintain absolute neutrophil counts or platelets counts above the required thresholds for study entry; use of erythropoietin stimulating agents and RBCs prior to study enrollment is allowed
* Neuropathy is a well described side effect of paclitaxel and carboplatin; patients may not have baseline peripheral neuropathy >= Grade 2
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain AT-101 tablets
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel within the last three months are excluded; subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would affect safety or limit compliance with study requirements
* Pregnant women are excluded from this study because the effects of AT-101 on the developing human fetus are unknown, but could potentially include teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AT-101, breastfeeding should be discontinued if the mother is treated with AT-101; these potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AT-101 or other agents used in this study; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with > grade 2 symptomatic hypercalcemia
* Patients with a myocardial infarction (MI) or cardiac (heart) surgery within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the highest dose level below the maximally administered dose at which no more than 1 out of 6 patients experience DLT graded according to NCI CTCAE version 4.0 | Up to 21 days

SECONDARY OUTCOMES:
AT-101 level (bound and unbound) | Up to 4 weeks after completion of study treatment
  Samples will be analyzed by validated LC-MS techniques.
Paclitaxel level (bound and unbound) | Up to 4 weeks after completion of study treatment
  Samples will be analyzed by validated LC-MS techniques.
Pharmacokinetics of AT-101 | Day 1 of courses 1 and 2 pre-AT-101 treatment and at 1, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, and 24 hours after AT-101 administration
  Pharmacokinetics will be determined by standard two-stage approaches using non-compartmental and compartmental modeling.
Pharmacokinetics of paclitaxel | Day 1 of courses 1 and 2 pre-AT-101 treatment and at 1, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, and 24 hours after AT-101 administration
  Pharmacokinetics will be determined by standard two-stage approaches using non-compartmental and compartmental modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Stein MN, Goodin S, Gounder M, Gibbon D, Moss R, Portal D, Lindquist D, Zhao Y, Takebe N, Tan A, Aisner J, Lin H, Ready N, Mehnert JM. A phase I study of AT-101, a BH3 mimetic, in combination with paclitaxel and carboplatin in solid tumors. Invest New Drugs. 2020 Jun;38(3):855-865. doi: 10.1007/s10637-019-00807-2. Epub 2019 Aug 6. PMID 31388792